CLINICAL TRIAL: NCT03890848
Title: Evaluation of the Effects of Home-based Functional Exercise on Patients With Anterior Cruciate Ligament Rupture Reconstruction Based on the Health Belief Model
Brief Title: Evaluation of the Effects of Home-based Functional Exercise on Patients With ACL
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: BMU2018MX030
Record Dates: First submitted 2019-03-11; First posted 2019-03-26 (Actual); Last update posted 2019-04-26 (Actual); Status verified 2019-04

CONDITIONS: Anterior Cruciate Ligament Rupture; Rehabilitation
Keywords: functional exercise; health belief model
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Wechat application intervention (Experimental): precautions and rehabilitation progress reminders and other news by optimized WeChat applet regularly
  Interventions: Behavioral: Wechat application reminder intervention
- routine guidance during discharge (Active Comparator): rehabilitation exercise guidance during routine discharge
  Interventions: Behavioral: routine guidance during discharge

INTERVENTIONS:
Behavioral: Wechat application reminder intervention — precautions and rehabilitation progress reminders and other news by optimized WeChat applet regularly
  Arms: Wechat application intervention
Behavioral: routine guidance during discharge — rehabilitation exercise guidance during routine discharge
  Arms: routine guidance during discharge

SUMMARY:
This study will evaluate the effect of home-based functional exercise on patients with anterior cruciate ligament rupture reconstruction based on the health belief model. About 360 participants will be randomly allocated into two groups. One group will randomized to receive precautions and rehabilitation progress reminders and other news by optimized WeChat applet regularly, while the other group will randomized to receive the rehabilitation exercise guidance during routine discharge.

DETAILED DESCRIPTION:
With the development of national fitness and sports, the incidence of anterior cruciate ligament (ACL) injuries has increased. ACL reconstruction is the best treatment for ACL injury. The success rate of surgery is high, but the patient still needs to rehabilitate after surgery, otherwise it is difficult to fully recover knee function. However, the rehabilitation medical resources in China are obviously insufficient. Patients who have undergone ACL reconstruction usually return home to work according to the rehabilitation plan. However, the adherence is still poor, and it is difficult to achieve the expected effect. The WeChat public account and its affiliated applets have been widely used in different health fields. The Health Belief Model (HBM) is a guiding theory commonly used in health education to guide patients for behavioral changes. This study aims to use the WeChat small program to explore the effects of optimized the existing Peking University Third Hospital Sports Medicine WeChat small program by using HBM to improve the adherence of patients with home-based functional exercise after ACL injury reconstruction.

ELIGIBILITY:
Inclusion Criteria:

* (1)Age between 18 and 45；
* (2)The first time to do simple ACL reconstruction, may be combined with cartilage -dressing and partial meniscectomy, patients with consistent postoperative rehabilitation plans;
* (3)Having the ability of Basic literacy, communication and accessibility;
* (4)Having a smartphone, using WeChat or can learn to use WeChat.

Exclusion Criteria:

* (1)Having history of joint infection, joint tuberculosis or osteomyelitis, or surgery in the lower extremities within 6 months;
* (2)Being combined with severe heart, brain, kidney and other organ dysfunction;
* (3)Having other serious knee injuries;
* (4)Being with mental illness or cognitive impairment, unable to learn and participate in rehabilitation training;
* (5)Having participated in other similar rehabilitation function training programs, or transferred to other medical institutions after discharge;
* (6)Doing not disagree to participate in the study,and not sign the informed consent.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 110 (Estimated)
Dates: Start 2019-04-01 (Actual); Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
qualified rate of knee joint activity | 6 weeks after surgery
  Knee joint activity reaches 125 degrees or above is judged to be qualified. Qualified rate is equal to the number of people who meet the standard divided by the total number in each group.
qualified rate of knee joint activity | 2 weeks after surgery
  Knee joint activity reaches 125 degrees or above is judged to be qualified. Qualified rate is equal to the number of people who meet the standard divided by the total number in each group.
qualified rate of knee joint activity | 12 weeks after surgery
  Knee joint activity reaches 125 degrees or above is judged to be qualified. Qualified rate is equal to the number of people who meet the standard divided by the total number in each group.

SECONDARY OUTCOMES:
Visual Analogue Scale | 2，6，12 weeks after surgery
  The Visual Analog or Analogue Scale (VAS) is designed to present to the respondent a rating scale with minimum constraints. Respondents mark the location on the 10-centimeter line corresponding to the amount of pain they experienced. This gives them the greatest freedom to choose their pain's exact intensity. It also gives the maximum opportunity for each respondent to express a personal response style. VAS data of this type is recorded as the number of millimeters from the left of the line with the range 0-100.
  1. Aitken, R. C. B. (1969). Measurement of feelings using visual analogue scales. Proceedings of the Royal Society of Medicine. 62, 989 - 993
  2. Freyd, M. (1923). The graphic rating scale. Journal of Educational Psychology, 43, 83 - 102
  3. Hayes, M. H. S. & D. G. Patterson (1921). Experimental development of the graphic rating method. Psychological Bulletin, 18, 98-99
SF-12 scale | 2，6，12 weeks after surgery
  The SF-12 scale is a simplified version of the Universal Concise Health-Related Quality of Life Scale SF-36 scale developed by the Boston Institute of Health Education. It includes 12 items and 8 dimensions for assessing physiological and psychological conditions.
  WARE J Jr，KOSINSKI M，KELLER S D.A 12-Item Short-Form Health Survey：construction of scales and preliminary tests of reliability and validity［J］．Med Care，1996，34（3）：220-233.
International Knee Documentation Committee (IKDC) Subjective Knee Form | 2，6，12 weeks after surgery
  International Knee Documentation Committee (IKDC) score: The IKDC score is divided into pain, stiffness, and difficulty in daily life. The score is 60. The lower the score, the better the knee function.
  van de Graaf, V. A., Wolterbeek, N., Scholtes, V. A. B., Mutsaerts, E. L. A. R., & Poolman, R. W. (2014). Reliability and Validity of the IKDC, KOOS, and WOMAC for Patients With Meniscal Injuries. The American Journal of Sports Medicine, 42(6), 1408-1416. https://doi.org/10.1177/0363546514524698

CONTACTS AND LOCATIONS:
Overall Officials: Yuping Yang, doctor, Study Director — Peking University Health Science Center
Locations (1):
- Peking University Third Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No